CLINICAL TRIAL: NCT00489307
Title: The Effect of Dexamethasone on Symptoms in Patients With Advanced Cancer
Brief Title: Dexamethasone for Symptom Burden in Advanced Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-0816; NCI-2012-01646 (Registry Identifier: NCI CTRP); MRSG-07-001-01-CCE (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors
Keywords: Advanced Cancer; Solid Tumors; Fatigue; Pain; Nausea; Anorexia; Dexamethasone; Decadron; Placebo
MeSH Terms: conditions — Fatigue; Pain; Nausea; Anorexia | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 4 mg orally two times a day for 14 days.
  On day 15 [ ± 3 days], all patients receive dexamethasone 4 mg orally twice a day for 7 days, and then the dose of dexamethasone tapered to 2 mg orally twice a day between days 22 to 28.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo by mouth (PO) twice daily for 14 days.
  On day 15 [ ± 3 days], all patients receive dexamethasone 4 mg orally twice a day for 7 days, and then the dose of dexamethasone tapered to 2 mg orally twice a day between days 22 to 28.
  Interventions: Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 4 mg PO (by mouth) twice daily x 14 days
  Other Names: Decadron
Drug: Placebo — Placebo PO twice daily x 14 days
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if dexamethasone can help to control symptoms such as fatigue, pain, nausea, weight loss, loss of appetite, sleep problems, and/or depression in patients with advanced cancer.

DETAILED DESCRIPTION:
Dexamethasone decreases inflammation and also suppresses the immune system.

If you are found to be eligible for this study, you will be randomly assigned (as in the toss of a coin) to receive either dexamethasone or a placebo by mouth in the morning and at night with food every day for 14 days. A placebo is a substance that looks like the study drug but which has no active ingredients. You will have an equal chance of being placed in either of the 2 groups. You, the medical staff, and researchers will not know to which group you have been assigned.

Beginning on Day 15 [± 3 days], regardless of if you were assigned to the dexamethasone or placebo group during the first 14 days, you will begin receiving the dexamethasone. On Days 15-21, you will receive dexamethasone 2 times a day. On Days 22-28 you will continue to take dexamethasone 2 times a day, but it will be at a lower dose level.

If you develop intolerable side effects while on this study, the medication will be stopped and you will be removed from the study.

You will be asked to return to the outpatient clinic on Days 8 [± 3 days], 15 [± 3 days] , 22 [± 3 days], and 29 [± 3 days] to answer a questionnaire about your cancer diagnosis, the medication you are taking, and the symptoms you are having (for example, pain, fatigue, nausea, appetite problems, sleep problems, depression, and your overall sense of well-being). The questionnaire will take approximately 30 minutes to complete. Blood (about 1 tablespoon) will be drawn to measure protein levels and to check the iron level in your blood. If you are unable to return to the clinic on days 8, 15, 22, or 29; the assessments will be done by the research nurse by phone; the blood work will not be done.

You will be considered off-study on Day 29 [ ± 3 days]. All study patients will have a 2 week follow-up on day 43 [± 3 days] after study drug has been discontinued, for safety and toxicity assessments. If you are unable to return to the clinic on day 43, the research nurse will do the safety and toxicity assessment by phone.

This is an investigational study. Dexamethasone has been approved by the FDA and is a commercially available drug. It is FDA approved at this dose level. Its use in this study, for this purpose, is investigational. About 160 patients will take part in this study. Up to 110 will be enrolled at the University of Texas (UT) MD Anderson Cancer Center. The other sites participating in this study are Lyndon Baines Johnson [LBJ] breast oncology clinic Houston Texas, and Four Seasons Hospice in Flat Rock, North Carolina.

ELIGIBILITY:
Inclusion Criteria:

1. Present with 3 or more symptoms during the last 24 hours (Pain, fatigue, chronic nausea, and anorexia/cachexia, sleep problems, depression or poor appetite), with an average intensity of >/= 4 on a 0-10 scale, in which 0= no symptom, and 10= worst possible symptom,
2. No clinical evidence of cognitive failure as evidenced by Memorial Delirium Assessment Scale (MDAS) score of 13 or less at baseline
3. Must be 18 years of older
4. No longer a candidate for aggressive anticancer therapy-such as receptor blockers (Iressa, etc.) Patients on oral or palliative chemotherapy are eligible for study if approved by primary oncologist prior to inclusion. Patients who are receiving IV chemotherapy are eligible for study if approved by primary oncologist and they have completed 1st line of chemotherapy and are deemed stable by primary oncologist. The PI of this study will obtain and document approval from the primary oncologist in the patient's study documents.
5. Life expectancy =/> 30 days
6. Must understand and sign written informed consent
7. Patients on topical, or inhaled corticosteroids are eligible for study. If patients have been on oral corticosteroids for </= 7 days prior to inclusion of study they are eligible for study.

Exclusion Criteria:

1. Allergy to Dexamethasone
2. Inability to complete the baseline assessment forms
3. Patients currently taking Megestrol, and not off drug for > 7 days
4. Anemia as defined as < 9 hemoglobin
5. Known history of human immunodeficiency virus (HIV)
6. Neutropenia as defined by an absolute neutrophil count (ANC) of < 1500 cells/mm
7. Patients with a history of diabetes will be excluded.
8. All major surgeries such as thoracotomy etc., that requires wound healing within last 2 weeks
9. Those who are currently receiving oral corticosteroid therapy or who have been on corticosteroid therapy >/= 8 days prior to study inclusion
10. Sepsis and/or acute, chronic, or ongoing infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-02-02 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2028-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced cancer with >= three Cancer related fatigue symptoms (ie, fatigue, pain, nausea, loss of appetite, depression, anxiety, or sleep disturbance) >= 4 of 10 on the Edmonton Symptom Assessment Scale (ESAS) were eligible.
Groups:
- Intervention Group (Dexamethasone): Dexamethasone 4 mg orally two times a day for 14 days.
- (Control Group) Placebo: Placebo by mouth (PO) twice daily for 14 days.
Period: Overall Study
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Started | 67 | 65
Completed | 43 | 41
Not Completed | 24 | 24
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Hospitalization unrelated to treatment | 10 | 7
Not completed — Surgery after assignment | 1 | 0
Not completed — Did not fill up the forms | 2 | 1
Not completed — Patient or family refusal | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo | Total
Number analyzed (Participants) | 67 | 65 | 132
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [29 to 89] | 60 [34 to 87] | 60 [29 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 28 | 70
  Male | 25 | 37 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 10 | 23
  White | 53 | 49 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 67 | 65 | 132
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) [Mean (Standard Deviation); unit: score on a scale] — FACIT Fatigue Subscale (13- item tool), FAACT Subscale (12-item tool) and FACIT-F Total Score (40-item tool). All of them asses self reported fatigue. All items in the above 3 tools are measured on a 4 point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The higher the score, the lower the fatigue level. FACIT Fatigue Subscale total score range is 0-52. FAACT Subscale total score range is 0-48. FACIT-F Total Score range is 0-160.
  score on a scale
    FACIT-F Subscale Score | 18.4 (10.47) | 21.57 (9.11) | 19.64 (9.98)
    FAACT Subscale score | 23.91 (8.28) | 25.69 (8.93) | 24.84 (8.58)
    FACIT_F- Total score | 88.66 (19.9) | 77.1 (23.83) | 80.85 (22.2)
Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: score on a scale] — The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. The total subscale score ranges from 0-21. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
  score on a scale
    HADS Anxiety score | 7.47 (4.18) | 7.46 (3.9) | 7.46 (4.03)
    HADS Depression score | 9.03 (5.72) | 4.22 (7.94) | 8.5 (3.8)
Edmonton Symptom Assessment System (ESAS) [Mean (Standard Deviation); unit: score on a scale] — The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity
  score on a scale
    ESAS Pain | 5.72 (2.43) | 5.14 (2.8) | 5.43 (2.63)
    ESAS Fatigue | 7.38 (1.89) | 5.14 (2.8) | 7.05 (1.89)
    ESAS Nausea | 2.64 (2.73) | 2.28 (2.76) | 2.46 (2.74)
    ESAS Depression | 3.13 (3.16) | 3.36 (3.11) | 3.24 (3.13)
    ESAS Anxiety | 3.64 (3.27) | 3.69 (2.91) | 3.66 (3.08)
    ESAS Drowsiness | 4.14 (3.19) | 4.2 (2.68) | 4.17 (2.94)

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Subscale Scores
Description: FACIT Fatigue Subscale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score range is from 0-52. The higher the score, the lower the fatigue level. It was measured as change in symptom score from Baseline to Day 15.
Time Frame: Baseline to Day 15
Population: A total of 48 participants were excluded from the analysis for various reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Number analyzed (Participants) | 43 | 41
score on a scale | 9 (10.3) | 3.1 (9.59)

2. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Pain
Description: ESAS was used to assess 10 symptoms commonly experienced by patients with cancer during the previous 24 hour. The severity of each symptom was rated on a numeric scale of 0 to 10 (0, no symptoms; 10, worst possible severity). Higher the score higher the severity of the symptom is. It was measured as change in symptom score from Baseline to Day 15.
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Number analyzed (Participants) | 43 | 41
score on a scale | -1.35 (3.11) | -0.17 (2.66)

3. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Nausea
Description: as for outcome 2
Time Frame: Baseline to Day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Number analyzed (Participants) | 43 | 41
score on a scale | -1.08 (2.95) | -0.36 (3.17)

4. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Appetite
Description: as for outcome 2
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Number analyzed (Participants) | 43 | 41
score on a scale | -2.19 (3.78) | -0.63 (3.11)

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Anxiety
Description: HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total range is from 0-21. The higher the score, the higher the severity of symptoms. It was measured as change in symptom score from Baseline to Day 15.
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Number analyzed (Participants) | 43 | 41
score on a scale | -0.66 (3.45) | -1 (3.54)

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Depression
Description: as for outcome 5
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
Number analyzed (Participants) | 43 | 41
score on a scale | -1.39 (3.59) | -0.31 (3.9)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 15
Description: Grading of adverse events as per National Cancer Institute Common Toxicity Criteria (version 3.0).
Arm/Group | Intervention Group (Dexamethasone) | (Control Group) Placebo
All-Cause Mortality (participants affected / at risk) | 1/43 | 1/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41
Other Adverse Events (participants affected / at risk) | 18/43 | 11/41
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Dexamethasone) (N=43) | (Control Group) Placebo (N=41)
Pain (Nervous system disorders) | 18 | 11
Insomnia (Nervous system disorders) | 3 | 6
Fatigue (Musculoskeletal and connective tissue disorders) | 8 | 6
Infection (General disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Edema (General disorders) | 1 | 4
Neuropathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 4
Nausea/Vomiting (Nervous system disorders) | 1 | 3
Blurred Vision (Nervous system disorders) | 1 | 0
Depression (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-04-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT00489307/Prot_SAP_000.pdf